CLINICAL TRIAL: NCT01071122
Title: A Prospective, Open-label, Active-controlled, Randomized Study Comparing Nifedipine GITS Versus Valsartan Versus a Combination of Both on Central Blood Pressure in Inadequately Controlled Essential Hypertension.
Brief Title: FOCUS (Nifedipine GITS's Effect on Central Pressure Assessed by Applanation Tonometry)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14696
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Central blood pressure; Nifedipine; Valsartan
MeSH Terms: conditions — Hypertension | interventions — Nifedipine; Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Nifedipine (Adalat, BAYA1040) and Valsartan
- Arm 2 (Active Comparator)
  Interventions: Drug: Nifedipine (Adalat, BAYA1040)
- Arm 3 (Active Comparator)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Nifedipine (Adalat, BAYA1040) and Valsartan — Combination treatment with nifedipine GITS 30mg and valsartan 80mg, Once daily
  Arms: Arm 1
Drug: Nifedipine (Adalat, BAYA1040) — Nifedipine 60mg, Once daily
  Arms: Arm 2
Drug: Valsartan — Valsartan 160mg, Once daily
  Arms: Arm 3

SUMMARY:
To determine whether the combination of nifedipine GITS and valsartan is more effective in reducing central blood pressure than nifedipine GITS or valsartan alone, and to determine whether nifedipine GITS is comparable to valsartan

ELIGIBILITY:
Inclusion Criteria:

* Untreated grade 2 or grade 3 hypertension defined by mean diastolic blood pressure (BP) >/= 100 and/or mean systolic BP >/= 160mmHg without anti-hypertensive treatment or Treated grade 2 hypertension defined by mean diastolic BP >/= 100 and/or mean systolic BP >/=160mmHg with current diuretics and/or beta-blockers use for >/= 4 weeks

Exclusion Criteria:

* Secondary form of hypertension
* Mean systolic BP >/= 200mmHg and or mean diastolic BP >/= 120mmHg
* Treated with other antihypertensive medication except diuretics or beta-blockers
* Type 1 diabetes mellitus
* Known cardiovascular disease including history of angina pectoris, heart failure, history of myocardial infarction or revascularization procedure, or cerebrovascular disease (including stroke and transient ischaemic attack) within the previous 12 months
* Renal insufficiency defined as a serum creatinine: >/= 1.7 mg/dl
* Pregnancy or not using contraceptive in childbearing aged women
* Breast feeding women
* Any disease or condition that in the opinion of the investigator may interfere with completion of the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Central systolic blood pressure | Week 8

SECONDARY OUTCOMES:
Change in central diastolic blood pressure and pulse pressure | Week 4,8
Change in central systolic blood pressure | Week 4
Change in brachial systolic blood pressure and diastolic blood pressure | Week 4,8
Change in brachial pulse pressure | Week4,8
Change in augmentation index and augmentation pressure | Week 4,8
Response rate(≥10 mmHg decrease of brachial SBP and ≥5mmHg decrease of brachial DBP) | Week 4,8
Control rate (≤140/90 mmHg, 130/80 mmHg for diabetes, of brachial BP | Week 4,8

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- South Korea (11):
  - Goyang, Gyeonggido
  - Goyang-si, Gyeonggido
  - Chungchungbuk-do, Korea
  - Seoul, Korea
  - Seoul, Seoul Teugbyeolsi
  - Busan
  - Gwangju
  - Joong-gu
  - Kungki-do
  - Seoul
  - Suwan

REFERENCES:
- [Derived] Park JB, Shin JH, Kim DS, Youn HJ, Park SW, Shim WJ, Park CG, Kim DW, Lee HY, Choi DJ, Rim SJ, Lee SY, Kim JH; FOCUS Investigators. Safety of the Up-titration of Nifedipine GITS and Valsartan or Low-dose Combination in Uncontrolled Hypertension: the FOCUS Study. Clin Ther. 2016 Apr;38(4):832-42. doi: 10.1016/j.clinthera.2016.02.025. Epub 2016 Mar 17. PMID 26996246